CLINICAL TRIAL: NCT05387785
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, 2-Period, 2-Arm, 4-Sequence, Crossover Phase 1b Study to Assess the Safety, Tolerability, and Pharmacokinetics of Ang-3070 in Subjects With Idiopathic Pulmonary Fibrosis Who Are Treatment-Naïve or Who Have Failed or Refused Standard of Care Treatment
Brief Title: Study to Assess the Safety and Tolerability of ANG-3070 in Subjects With Idiopathic Pulmonary Fibrosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Angion Biomedica Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ANG3070-IPF-102
Record Dates: First submitted 2022-05-17; First posted 2022-05-24 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, double-blind, placebo-controlled, cross-over design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 500 mg QD (Experimental): 500 mg QD of ANG-3070 will be taken once a day for 10 days.
  Interventions: Drug: ANG-3070
- 300 mg BID (Experimental): 300 mg BID of ANG-3070 will be taken twice a day for 10 days.
  Interventions: Drug: ANG-3070
- Placebo-to-match 500 mg QD (Placebo Comparator): Placebo-to-match 500 mg QD of ANG-3070 will be taken once a day for 10 days.
  Interventions: Drug: Placebo
- Placebo-to-match 300 mg BID (Placebo Comparator): Placebo-to-match 300 mg BID of ANG-3070 will be taken twice a day for 10 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ANG-3070 — Orally administered tyrosine kinase inhibitor capsule.
  Arms: 300 mg BID; 500 mg QD
Drug: Placebo — Orally administered placebo capsule
  Arms: Placebo-to-match 300 mg BID; Placebo-to-match 500 mg QD

SUMMARY:
The purpose of this study is to assess safety and tolerability of once daily (QD) and twice daily (BID) dosing of ANG-3070 in subjects with idiopathic pulmonary fibrosis (IPF) who are treatment-naïve, refused therapy, or discontinued for any reason current standard of care with nintedanib or pirfenidone.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be willing and of sufficient mental capacity to give written informed consent and comprehend the importance of adhering to study treatment and requirements.
2. Male or female subjects aged 40 years and older at the time of informed consent.
3. Substantiated diagnosis of IPF based on clinical, radiological, and/or pathologic data to the exclusion of alternate diagnoses that would contribute to extant interstitial lung disease (ILD) based on the opinion of the subject's physician using current diagnostic criteria.
4. Subject:

   * Is naïve to therapy with nintedanib or pirfenidone OR
   * Refuses therapy with nintedanib or pirfenidone OR
   * Had nintedanib or pirfenidone discontinued due to any reason, 4-week washout required

Exclusion Criteria:

1. Diagnosis of asthma or chronic obstructive pulmonary disease (COPD).
2. Current tobacco use (quit at least 1 month prior to study for inclusion).
3. Presence of active infection requiring ongoing therapy with systemic antibiotics and/or antivirals.
4. Diagnosis of connective tissue disease.
5. Known cause of ILD diagnosed.
6. Active malignancy aside from local carcinoma.
7. AST or ALT or total bilirubin > 2x upper limit of normal (ULN).
8. Pregnancy and/or lactation; positive serum beta human chorionic gonadotropin (β-HCG) during screening.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of the frequency and severity of treatment-emergent adverse events (TEAEs), including clinically significant abnormal findings from vital signs. | Period 1 Day 1 and Day 30
Change from baseline of the frequency and severity of treatment-emergent adverse events (TEAEs), including clinically significant abnormal findings from 12-lead electrocardiograms (ECGs). | Period 1 Day 1 and Day 30
Change from baseline of the frequency and severity of treatment-emergent adverse events (TEAEs), including clinically significant abnormal findings from laboratory test results. | Period 1 Day 1 and Day 30
Change from baseline of the frequency and severity of treatment-emergent adverse events (TEAEs), including clinically significant abnormal findings from physical examination. | Period 1 Day 1 and Period 2 Day 1